CLINICAL TRIAL: NCT04125277
Title: SONImage Study: Can Molecular Imaging Predict Outcome to First-line Endocrine Treatment ± CDK 4/6 Inhibition in Advanced ER+ Breast Cancer
Brief Title: The SONImage Study
Acronym: SONImage
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other); BOOG Study Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M22SIM
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imaging (Experimental): One visit to either the UMCG or Amsterdam UMC-location VUMC is required for the FES-PET scan, and possibly one additional visit for an FDG-PET. A FES- or FDG-PET scan plus low dose CT will each induce an extra radiation burden of about 6.1 mSv (210 MBq injected for an average patient of 70 kilogram body weight).
  Interventions: Other: FES-PET scan, and possibly one additional visit for an FDG-PET

INTERVENTIONS:
Other: FES-PET scan, and possibly one additional visit for an FDG-PET — One visit to either the UMCG or Amsterdam UMC-location VUMC is required for the FES-PET scan, and possibly one additional visit for an FDG-PET. A FES- or FDG-PET scan plus low dose CT will each induce an extra radiation burden of about 6.1 mSv (210 MBq injected for an average patient of 70 kilogram body weight).

SUMMARY:
SONImage is a multicenter prospective imaging side study, in which a baseline FES-PET is added to conventional work up, in 100 patients with ER+ MBC who will receive endocrine treatment ± CDK 4/6 inhibition within the SONIA study (NCT03425838). SONImage will be executed in two Dutch centers: UMCG and Amsterdam UMC-location VUMC. The aim of the SONImage study is to (1) assess the relationship between FES/FDG-PET heterogeneity patterns at baseline and PFS for first-line endocrine treatment ± CDK 4/6 inhibition in ER+ MBC, and (2) to further improve that by developing a prediction model, within the SONIA study. This molecular imaging based multivariable prediction model may provide a unique measure of benefit of adding CDK 4/6 inhibition to first-line endocrine treatment, allowing patients and providers to weigh individual benefits and (long term) burden for optimized treatment decisions.

DETAILED DESCRIPTION:
Estrogen receptor positive (ER+) breast cancer is the most common cancer and the most frequent cause of cancer-related death in women in the Western World. Cyclin-dependent kinase 4 and 6 (CDK 4/6) inhibitors improve outcome, when added to standard first- and second-line endocrine therapy. However, they also add patient- and financial burden due to (long term) increased toxicity and hospital visits. Therefore, benefits of additional CDK 4/6 inhibitors should be weighed against their burden. Tools to support such treatment decisions by patients and providers are currently lacking. Whole body heterogeneity of ER expression, measured by 16α-[18F]fluoro-17β-estradiol (FES)-PET scan and 18F-fluorodeoxyglucose (FDG)-PET scan was related to time to progression on combined treatment in previous work. Therefore in SONImage a baseline FES-PET is added to conventional work up, in 100 patients with ER+ MBC who will receive first line endocrine treatment ± CDK 4/6 inhibition within the SONIA study. The objectives are 1. to correlate PFS1 (according to SONIA criteria) to baseline FES/FDG-PET heterogeneity; 2. to assess interaction between baseline FES/FDG-PET heterogeneity, treatment allocation, and PFS1 (according to SONIA criteria); 3. to correlate response measurements of individual lesions to baseline FES/FDG heterogeneity and detailed FES/FDG imaging features; 4. to develop a multivariable model to predict individual PFS benefit to first-line AI ± CDK 4/6 inhibition, based on detailed FES/FDG image features and standard clinicopathological information, in n=100 SONIA patients; 5. to validate this prediction model in two independent patient cohorts with baseline FES/FDG-PET scans (Dutch IMPACT-MBC trial; international ET-TRANSCAN trial). This molecular imaging based multivariable prediction model may provide a unique measure of benefit of adding CDK 4/6 inhibition to first-line endocrine treatment, allowing patients and providers to weigh individual benefits and (long term) burden for optimized treatment decisions. Particularly for the approximately 25% of patients with ER+ MBC who have an excellent- or poor outcome despite CDK 4/6 inhibition in the first-line, this could have profound implications, as they may refrain from combined treatment. Ultimately, this could potentially contribute to FES/FDG-PET based treatment decisions in clinical practice, reduction of unnecessary toxicity and costs, while improving patient outcome and QoL.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is eligible and participates in the SONIA trial for ER+ MBC.
2. Able to give written informed consent and to comply with the SONImage protocol.
3. Documentation of histologically confirmed diagnosis of estrogen receptor (ER) expression >10% breast cancer based on local results. The receptor status can be determined on the primary tumor or on a tumor biopsy of a metastatic lesion.

Exclusion Criteria:

1. A patient who meets the exclusion criteria of the SONIA trial (see SONIA protocol).
2. Contra-indication for PET imaging.
3. Use of estrogen receptor ligands (i.e. tamoxifen or fulvestrant) ≤ 5 weeks before FES-PET imaging.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival after first line treatment (PFS1) | 5 years
  Progression-free survival after first line treatment (PFS1) defined as time from randomization until objective disease progression, symptomatic deterioration, or initiation of a new therapeutic agent on first line treatment, death, or progression during a break in initial therapy and without further therapy within one month, whichever occurs first.

SECONDARY OUTCOMES:
Patient response | 5 years
  Per patient response according to RECIST1.1
Response measurement individual lesion | 5 years
  Change in size (=response measurement) per individual lesion at the largest measurable response measured on CT compared to baseline CT
Response measurement target lesions | 5 years
  - Per patient trajectory of change in size of target lesions according to RECIST 1.1, from baseline CT until CT at progression of disease.

OTHER OUTCOMES:
Association baseline FES/FDG-PET heterogeneity score with primary endpoint. | 5 years
  Cox-regression to estimate HRs for PFS and corresponding 95% CIs between FES/FDG heterogeneity groups, while adjusting for treatment allocation.

CONTACTS AND LOCATIONS:
Overall Officials: C. P. Schröder, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (2):
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - VU Medical Center, Amsterdam